CLINICAL TRIAL: NCT05975502
Title: Congenital Syphilis in Switzerland: a National Multicentric Retrospective Epidemiological Study
Brief Title: Congenital Syphilis in Switzerland
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Fonds national Suisse (Unknown)
Responsible Party: Principal Investigator, Laurence Toutous Trellu, Medical Doctor, University Hospital, Geneva
Other Study IDs: Study 2022-01296
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Congenital Syphilis
Keywords: Congenital syphilis; pregnant women with syphilis
MeSH Terms: conditions — Syphilis, Congenital | interventions — Epidemiologic Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with positive syphilis serology: Pregnant women with blood TPHA/TPPA ≥ 80
  Interventions: Other: Epidemiological study
- Children born with positive syphilis serology: Children born from mothers with syphilis during pregnancy and / or with blood TPHA/TPPA ≥ 80 at birth
  Interventions: Other: Epidemiological study

INTERVENTIONS:
Other: Epidemiological study — Study of epidemiological characteristics of women with syphilis during pregnancy and of children born from mothers with syphilis during pregnancy.

SUMMARY:
A retrospective national epidemiological Swiss study was conducted to establish a real prevalence and description of congenital syphilis, and to better classify the reported congenital syphilis.

Maternal risk factors to contract syphilis (i.e. socio-demographic, cultural and clinical factors) were also evaluated, in order to focus on prevention of these targeted population.

Follow up of the children born from mother with syphilis during pregnancy, until age 6, was recorded to evaluate the risk of congenital syphilis following treatment of maternal syphilis.

DETAILED DESCRIPTION:
We conducted an observational and descriptive retrospective multicentric national study in Switzerland of all pregnant women diagnosed with syphilis during their pregnancy and their babies from childbirth to age 6.

Retrospective clinical and biological data already collected in the patient's medical file from 2012 until 2021 were collected from pregnant women diagnosed with syphilis during their pregnancy and their babies from childbirth to age 6, in Swiss universities and cantonal hospitals.

Cases were collected through the computerized laboratory records by selecting all pregnant women with a positive TPHA / TPPA serology and children born to mothers who had syphilis diagnosed during pregnancy or / and with a positive TPHA / TPPA serology. Data collected included clinical information's, results of biological tests and imagery available from the hospital's internal archiving system and registered on two standardized coded case report forms (one for the mother and one for the babies).

Recent guidelines from the Centers for Disease Control recommend testing for syphilis at the first prenatal visit and again at 28 weeks gestation and at delivery if at high risk for syphilis acquisition during pregnancy. The identification, through the collection of epidemiological data, of risk factors for developing congenital syphilis during pregnancy may improve the prevention of congenital syphilis in the population at risk. It would make it possible to carry out preventive actions, repeated screening of syphilis during pregnancy and closer monitoring in a targeted population of women of childbearing age.

Thus, a proactive sentinel network could be developed to limit new cases of congenital syphilis in Switzerland, with the development of tools that could send alerts to the various specialists involved (biologist, gynaecologist, paediatrician, dermatologist) when a syphilis serology comes back positive in a pregnant woman.

This project is part of one of WHO's goals to eradicate congenital syphilis, as a better knowledge of congenital syphilis could lead us to propose solutions intended to reduce this serious disease. All the more that congenital syphilis is preventable by syphilis pregnancy screening and the burden of congenital syphilis is avoidable with a simple cost-effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who had a positive TPHA / TPPA serology during pregnancy.
* All children born to mothers who had syphilis diagnosed during pregnancy or / and with a positive TPHA / TPPA serology.

Exclusion Criteria:

* Document in the medical file attesting to a refusal of consent to the re-use of the data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women with a positive syphilis screening and their babies until age 6 from university and cantonal hospitals in Switzerland (Geneva, Lausanne, Zurich, Bern, Basel, Saint Gallen, Valais, Lugano) in dermatology, paediatric and gynaecology wards.
  Retrospective analysis of data from medical records.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
To quantify the number of syphilis cases during pregnancy and the number of congenital syphilis cases. | Ten years: 2012 - 2021
  Study of medical records of all university hospitals in Switzerland through a national observational epidemiological study from 2012 until now.
To describe maternal characteristics associated with congenital syphilis (i.e. socio-demographic, cultural and clinical factors), in order to focus on prevention of these targeted population. | Ten years: 2012 - 2021
  Study of medical records of all university hospitals in Switzerland through a national observational epidemiological study from 2012 until now.

SECONDARY OUTCOMES:
To describe the clinical itinerary, follow-up and development of their baby from birth to age 6. | Ten years: 2012 - 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Laurence Toutous Trellu, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kimball A, Bowen VB, Miele K, Weinstock H, Thorpe P, Bachmann L, McDonald R, Machefsky A, Torrone E. Congenital Syphilis Diagnosed Beyond the Neonatal Period in the United States: 2014-2018. Pediatrics. 2021 Sep;148(3):e2020049080. doi: 10.1542/peds.2020-049080. PMID 34465590
- [Background] Salome S, Cambriglia MD, Scarano SM, Capone E, Betts I, Pacella D, Sansone M, Mazzarelli LL, Lo Vecchio A, Ranucci G, Marinosci GZ, Capasso L, Salvatore P, Raimondi F. Congenital syphilis in the twenty-first century: an area-based study. Eur J Pediatr. 2023 Jan;182(1):41-51. doi: 10.1007/s00431-022-04703-5. Epub 2022 Nov 14. PMID 36376519
- [Background] Townsend CL, Francis K, Peckham CS, Tookey PA. Syphilis screening in pregnancy in the United Kingdom, 2010-2011: a national surveillance study. BJOG. 2017 Jan;124(1):79-86. doi: 10.1111/1471-0528.14053. Epub 2016 May 24. PMID 27219027
- [Derived] Alberto C, Wagner N, Fougere Y, Meyer Sauteur PM, Scherler G, Aebbi-Popp K, Baumann M, Schobi N, Catho G, Emonet S, Polli C, Kottanattu L, Kahlert C, Baud D, Coste A, Martinez De Tejada B, Posfay Barbe KM, Toutous Trellu L. Syphilis in pregnant women and congenital syphilis from 2012 to 2021 in Switzerland: a multicentre, retrospective study. Swiss Med Wkly. 2024 Nov 1;154:3678. doi: 10.57187/s.3678. PMID 39509430
- See also: Syphilis and congenital syphilis in Europe - A review of epidemiological trends (2007-2018) and options for response — https://www.ecdc.europa.eu/en/publications-data/syphilis-and-congenital-syphilis-europe-review-epidemiological-trends-2007-2018
- See also: World Health Organisation - Governance guidance for the validation of elimination of mother-to-child transmission of HIV and syphilis — https://www.who.int/publications-detail-redirect/governance-guidance-for-validation-of-emtct-syphilis-hiv
- See also: Office fédéral de la santé publique. - Chiffres Maladies infectieuses - Syphilis — https://www.bag.admin.ch/bag/fr/home/zahlen-und-statistiken/zahlen-zu-infektionskrankheiten.html